CLINICAL TRIAL: NCT01369823
Title: Prospective, Multicenter, Non-interventional Post Market Release Study , to Examine Whether Pump Treatment Combined With the Use of Continuous Glucose Monitoring System is a Mean to Normalize Glycaemic Control.
Brief Title: Diabetes Multicenter Observational Study (DIAMOND-1-)
Acronym: DIAMOND-1
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Medtronic Hellas Medical Devices ΑEE (Industry)
Responsible Party: Dr. Eleni Papavasileiou / Field Clinical research Specialist, Medtronic Hellas Medical Devices ΑEE
Other Study IDs: Version 1.0 - 12/Sep/2008
Record Dates: First submitted 2011-06-07; First posted 2011-06-09 (Estimated); Last update posted 2011-06-09 (Estimated); Status verified 2011-06

CONDITIONS: Diabetes
Keywords: HbA1c; Paradigm 522/722 Infusion Pump; Transmitter (MMT-7703WW); Sensor MMT-7002 (i.e. Glucose Sensor); Levels of HbA1c at enrollment higher than 7
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to examine whether pump treatment combined with the use of continuous glucose monitoring system is a mena to normalize glycaemic control.

DETAILED DESCRIPTION:
In this study, 100 subjects, users of Paradigm 522/722 Infusion Pump and Self- Monitoring Blood Glucose finger sticks for the control of their glucose levels for at least 3 months prior enrollment will participate. Moreover the subjects won't have achieved the best blood glucose control, with an average HbA1c above 7% and should meet all the inclusion and none of the exclusion criteria. The HbA1c value for screening purposes can be taken from the medical chart, while in the enrollment visit according to current medical practice of each investigational center, the sample taken for HbA1c measurement will be analyzed centrally by HPLC, in a lab in Germany. In all enrolled patients a continuous glucose monitoring system will be provided. Since this is an observational study, the provision of the glucose monitoring system will be based on medical justification and will not be done per protocol requirement. All subjects will be followed for 3 months according to the current medical practice of each investigational center. All other visits, e.g. patient comes into the hospital because of symptoms, will also be recorded as unscheduled visits. These visits are usually linked to Adverse Events.

ELIGIBILITY:
Inclusion Criteria:

* Subjects and/or their legal representative must sign the Patient Data Release Form (PDRF).
* Subjects must be aged between 12 and 45 years old.
* Subjects must be pump and Self- Monitoring Blood Glucose fingersticks users for at least 3 months and no more than 9 months.
* HbA1c >7.0% with a measurement no older than three months prior to enrollment.
* Diagnosed T1D at least 1 year before study entry.
* Subjects must be able to understand how to use the Paradigm REAL-Time System and how to adjust and administer corrective treatment.
* Subjects should not have used the sensor in the past.

Exclusion Criteria:

* Hearing or vision impairment so that alarms can not be recognized.
* Alcohol or drug abuse other than nicotine.
* Subjects suffering from severe chronic disease or genetic disorder other than T1D. (i.e. Down syndrome etc.)
* Subjects suffering from allergy.
* Subjects in pregnancy or with desire to conceive during study.
* Subjects participating in other device or drug studies.

Ages: 12 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: This is an observational pilot study that does not have a statistically powered primary hypothesis. The data collected during this study are for the purpose of accumulating information that may generate research ideas and lead to publications. For this reason a sample size of 100 subjects has been defined. The statistical analysis will be descriptive statistics and will be described in a separate statistical analysis plan. Moreover any enrolled patient that has a sensor usage % in the end of the study that is less than 65% will be excluded from the analysis.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2009-06; Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
The levels of HbA1c will be investigated on patients combining the pump therapy with continuous glucose monitoring over a period of three months. | 2 years

SECONDARY OUTCOMES:
To evaluate the impact of continuous sensing on the variability of glucose | 2 years
To examine the frequency of hypoglycemic events. | 2 years
To examine the frequency of ketoacidosis events | 2 years
To examine the frequency of Emergency Department visits | 2 years
To examine the frequency of hospitalizations | 2 years
To examine the duration of hospitalizations | 2 years
To evaluate the daily insulin requirements | 2 years
To evaluate the % sensor usage | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Charalampos Vasilopoulos, Dr., Principal Investigator — General Hospital of Athens "Evaggelismos"; Christos Zoupas, Dr., Principal Investigator — Diagnostic and Therapeutic Center of Athens "Hygeia"; Marriana Benroubi, Dr., Principal Investigator — General Hospital of Athens "POLICLINIC"; Christina Kanaka, Dr., Principal Investigator — Children General Hospital " Agia Sofia"; Nikolaos Tentolouris, Dr., Principal Investigator — General Hospital of Athens "LAIKO"; Maria Alevizaki, Assoc. Prof., Principal Investigator — General Hospital of Athens "ALEXANDRA"; Andrianni Gerasimidi, Dr., Principal Investigator — Children Hospital "Aglaia Kiriakou"; Andreas Melidonis, Dr., Principal Investigator — General Hospital of Peiraeus "TZANEIO"; Dimitrios Mamoulakis, Dr., Principal Investigator — University Hospital of Heraklion; Angelos Pappas, Dr., Principal Investigator — "Venizeleio - Pananeio" General Hospital of Heraklion; Triantafillos Didaggelos, Lecturer, Principal Investigator — University Hospital of Thessalonica " AXEPA",Α' Propedeutic Pathology Clinic; Ioannis Giovos, Assoc. Prof., Principal Investigator — University Hospital of Thessalonica " AXEPA" ,Α' Pathology Clinic; Emmanouil Pagkalos, Dr., Principal Investigator — General University Hospital of Thessalonica "PAPAGEORGIOU",Α' Pathology Clinic; Asimina Galli, Ass. Prof., Principal Investigator — General University Hospital of Thessalonica "PAPAGEORGIOU",D' Pediatric Clinic; Christos Manes, Dr., Principal Investigator — General University Hospital of Thessalonica "PAPAGEORGIOU",Β' Pathology Clinic; Agathoklis Tsatsoulis, Prof., Principal Investigator — General University Hospital of Ioannina; Ioannis Chabeos, Lecturer, Principal Investigator — General University Hospital of Rio- Patra